CLINICAL TRIAL: NCT02678585
Title: Nalbuphine as an Adjuvant to Intravenous Regional Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Bakri, Associate professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 000087161
Record Dates: First submitted 2016-02-04; First posted 2016-02-10 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Nalbuphine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Nalbuphine (Active Comparator): 53 patients received intravenous regional lidocaine plus Nalbuphine
  Interventions: Drug: Nalbuphine
- Control group (Other): 53 patients received intravenous regional lidocaine
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Nalbuphine — 53 patients received intravenous regional lidocaine plus nalbuphine
  Arms: Nalbuphine
Drug: Lidocaine — 53 patients received intravenous regional lidocaine
  Arms: Control group

SUMMARY:
The effect of addition of nalbuphine to lidocaine in intravenous regional anesthesia

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* American Society of Anesthesiologists (ASA) physical status I-II
* age between 20 and 50 years old
* scheduled for elective unilateral short hand surgery

Exclusion Criteria:

* allergy to study medications
* body mass index > 35 kg/m2
* patients with sickle cell disease or Reynaud disease
* patient refusal

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Tourniquet and postoperative pain measured by visual analogue scale | 4 hours

SECONDARY OUTCOMES:
Cortisol level | 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt